CLINICAL TRIAL: NCT01752608
Title: A Randomized, Comparator-Controlled, Two-Arm, Parallel Group Study to Determine the Safety and Efficacy of eCBT Mood®, a Handheld, Computerized, Electronic Cognitive Behavioral Therapy Application, in Patients With Major Depressive Disorder
Brief Title: Efficacy of Electronic Cognitive Behavioral Therapy Application to Treat Major Depressive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: MindApps (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eCBT 201
Record Dates: First submitted 2012-12-16; First posted 2012-12-19 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Real-time; iPhone; CBT; Cognitive behavioral therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- eCBT Mood (Experimental): Electronic cognitive behavioral therapy application running on the iPhone and iPod Touch.
  Interventions: Behavioral: eCBT Mood
- Mood Tracker (No Intervention): Mood monitoring application running on the iPhone and iPod Touch

INTERVENTIONS:
Behavioral: eCBT Mood — A handheld, computerized, electronic cognitive behavioral therapy (CBT) application
  Arms: eCBT Mood

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of an electronic cognitive behavioral therapy application (eCBT Mood) compared to a control group consisting of a mood monitoring handheld computer application in the treatment of patients with mild to moderate major depressive disorder.

DETAILED DESCRIPTION:
This is a prospective, randomized, comparator-controlled, two-arm, parallel group study to examine the safety and efficacy of eCBT Mood, a handheld, computerized, electronic cognitive behavioral therapy (CBT) application, in patients with major depressive disorder (MDD). The study will involve 100 patients with mild to moderate MDD randomly assigned to daily use of either a CBT application focused on depression ('eCBT Mood'; MindApps, llc) or a comparator-controlled group using a mood monitoring application ('Mood Tracker'; GP International). This study design and duration of the study is consistent with other studies employing comparator-controlled designs in the study of CBT interventions, including computerized CBT interventions, among patients with MDD (e.g., Andrews et al., 2010; McKendree-Smith et al., 2003).

After being screened to ensure that the patients meet the required diagnostic, depression severity, and other inclusion criteria, patients will be randomly assigned (1:1) to use either eCBT Mood, a computer application running on the Apple® iPhone™ or iPod Touch® handheld computer platforms. The application includes: (1) a psychoeducation module on the relationships among thoughts, feelings, and behaviors, (2) a 6-item daily depression assessment with the option to e-mail the summary score and suicidal ideation assessment response to a 3rd party, (3) a negative automatic thought identification module, (4) a feelings and thoughts log, (5) a module enabling the user to challenge their negative automatic thoughts, (6) an assessment and challenge module regarding core beliefs which underlie many automatic thoughts, (7) optional compliance reminders to use the application or take medicines, and (8) links to behavioral science-based online content regarding MDD from PsychCentral (see www.psychcentral.com). In contrast, the comparator control condition will use Mood Tracker, which is also a a computer application running on the Apple iPhone or iPod Touch handheld computer platforms. This application enables users to rate their mood using expressive faces on a daily basis, log about their daily feelings, and also has an option enabling an e-mail to be sent to a 3rd party regarding their daily mood ratings.

Throughout the 8-week study period, patients will complete both in-person and telephone-based assessments of their depression severity, mood, frequency of negative automatic thoughts, and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 65 at the date of consent.
* Diagnosis of MDD consistent with the DSM-IV-TR as assessment by the Mini International Neuropsychiatric Interview (MINI).
* Owns and has access to an iPhone or iPod Touch capable of downloading and running either eCBT or the comparator mood monitoring application.
* At the screening and visits, must exhibit mild to moderate MDD with scores between 17 and 34 on the MADRS, inclusive. Subjects with scores >34 on the MADRS will be referred by the Study Investigator for alternative psychotherapeutic and/or pharmacological care for their depression.
* Note that no subjects are to be discontinued from any pharmacotherapies used to treat depression solely for the purpose of qualifying for this study. Be willing and able to refrain from the following therapies for the duration of the study:
* All approved pharmacotherapies for MDD, including serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, monoamine oxidase inhibitors, tricyclic and tetracyclic antidepressants, bupropion, mood stabilizers, and adjunctive antipsychotics.
* Medical device therapies for depression, including transcranial magnetic stimulation, vagal stimulation, electroconvulsive shock therapy, and others.
* Beginning any type of group or individual psychotherapy.
* Beginning another clinical trial for major depressive disorder or other condition.
* Patients' primary language must be English.
* Subject is willing and has an understanding and ability to fully comply with study procedures and restrictions defined in this protocol.

Exclusion Criteria:

* Depression severity, as measured by either:
* Clinician judgment that the patient's depression is too severe to make self-help resource a viable treatment option.
* Depression severity as measured by a scores >34 on the MADRS.
* Clinician assessed high risk of suicide or self-harm.
* Intellectual disability or physical limitation that would prevent use of the computerized handheld intervention.
* Comorbid psychopathology where the primary disorder is not depression.
* Within the past 3 months has had a course of treatment with psychotherapy or pharmacotherapy for depression.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Change from baseline to Week 8

SECONDARY OUTCOMES:
Automatic Thoughts Questionnaire-Revised (ATQ-R) | Change from baseline to Week 8
Beck Depression Inventory, 2nd Edition | Change from baseline to Week 8
Profile of Mood States, Short-Form (POMS-SF) | Change from baseline to Week 8

OTHER OUTCOMES:
Adverse events | As assessed at each of 9 visits over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hufford, Phd, Study Chair — CEO of MindApps
Locations (2):
- United States (2):
  - Compass Research, LLC: North Clinic, Leesburg, Florida
  - Compass Research LLC, Orlando, Florida